CLINICAL TRIAL: NCT04452591
Title: A Phase 3 Study of Cretostimogene Grenadenorepvec in Patients With Non-Muscle Invasive Bladder Cancer (NMIBC) Unresponsive to Bacillus-Calmette-Guerin (BCG)
Brief Title: Study of Cretostimogene Given in Patients With Non-Muscle Invasive Bladder Cancer ,Unresponsive to Bacillus-Calmette-Guerin
Acronym: BOND-003
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CG Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG3002S
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Non Muscle Invasive Bladder Cancer; High-grade Ta/ T1 Papillary Disease Bladder Cancer
Keywords: high-grade Ta papillary disease; high-grade T1 papillary disease; carcinoma in situ; Bacillus-Calmette-Guerin unresponsive
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ | interventions — dodecyl maltoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort C(All Countries):Enrollment Closed (Experimental): Patients with CIS with or without HG Ta/T1 papillary disease. Cretostimogene will be administered intravesically following a series of bladder washes with 5% DDM and normal saline. Cretostimogene will be administered weekly x 6 on Weeks 1, 2, 3, 4, 5, and 6. If the patient has disease recurrence at Week 13, they will receive another cycle of 6 weekly treatments. If there is no disease present at Week 13 then the patient will receive 3 weekly treatments. Cohort C(All Countries):Beginning at Week 25, patients will receive weekly x 3 treatments every 12 weeks through week 51 then every 6 months and then a last treatment at Weeks 73, 74, and 75 until the tumor returns or study treatment is completed at Week 97. Cohort C Extension( Japan and the US) At Week 25, patients will receive weekly x 3 treatments every 12 weeks through week 51 then every 6 months starting at Weeks 73, 74, and 75 through Weeks 157, 158, and 159 until the tumor returns or study treatment is completed at Week 159.
  Interventions: Biological: Cretostimogene Grenadenorepvec; Other: n-dodecyl-B-D-maltoside
- Cohort P(Japan and United States Only) :Open to Enrollment (Experimental): HG Ta/T1 papillary disease bladder cancer patients.
  In Cohort P, cretostimogene will be administered at a dose of 1 × 1012vp IVE following instillation of 5% DDM. Cretostimogene will be administered every week for 6 treatments on Weeks 1, 2, 3, 4, 5, and 6. If the patient has recurrence at Week 13 or any timepoint, the patient will receive a second induction of 6 weekly treatments (Weeks 13, 14, 15, 16, 17, and 18.). If the tumor has not returned they will receive 3 weekly treatments every 12 weeks (approximately 3 months) starting Weeks 13, 14, and 15 through Week 51 (approximately 12 months), and then every 6 months starting at Weeks 73, 74, and 75 (approximately 18 months) through Month 36.
  Interventions: Biological: Cretostimogene Grenadenorepvec; Other: n-dodecyl-B-D-maltoside

INTERVENTIONS:
Biological: Cretostimogene Grenadenorepvec — Engineered Oncolytic Adenovirus
Other: n-dodecyl-B-D-maltoside — Transduction-enhancing agent.
  Other Names: DDM

SUMMARY:
This is a Phase 3, open-label, single arm trial designed to evaluate Cretostimogene patients with NMIBC who have failed prior BCG therapy. Up to approximately 115 CIS bladder cancer patients with or without HG Ta or HG T1 papillary disease will be enrolled under the original protocol through Amendment 4, which will comprise Cohort C. Cohort C is closed to enrollment.

Under Amendment 5-1, Cohort P was added to enroll up to 70 patients with HG Ta/T1 papillary bladder cancer.

Under Amendment 6, the target number of patients enrolled in Cohort P was increased to 75. Cohort P is open to enrollment

Cohort C and Cohort P will be analyzed and reported separately. Patients will have had to fail prior BCG therapy which is defined as having persistent or recurrent disease within 12 months (Cohort C) or 6 months (Cohort P) following the completion of adequate BCG therapy for HGUC

DETAILED DESCRIPTION:
Cohort C(All Countries) :

An open-label trial designed to evaluate Cretostimogene + DDM in patients with NMIBC who have failed prior BCG therapy. Single treatment arm that enrolled 115 patients with carcinoma in situ with or without concomitant high-grade Ta or T1 papillary disease

BCG failure is defined as a persistent or recurrent disease within 12 months of completion of adequate BCG therapy.

Cohort P(Japan and the United States Only):

To determine the all-cause High Grade Event Free Survival (HG-EFS) of cretostimogene in up to 75 patients with BCG-unresponsive HG Ta/T1 papillary disease without CIS.

BCG failure is defined as a persistent or recurrent disease within 6 months of completion of adequate BCG therapy.

ELIGIBILITY:
Cohort C Inclusion Criteria

In order to be eligible for participation in this trial, the patient must:

* Be ≥18 years of age (or legal age of majority in the jurisdiction) on day of signing informed consent.
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Have pathologically confirmed (WHO grading system employed for tumor grading) (Compérat 2019) BCG unresponsive CIS. Patients with BCG unresponsive CIS are those unlikely to benefit from, and who will not be receiving, further intravesical BCG. There is no maximum limit to the amount of prior BCG treatment, but maintenance BCG should be administered on a schedule consistent with standard induction-maintenance protocols (e.g., BCG weekly × 6 then weekly × 3 weeks administered at Months 3, 6, 12, 18, 24, and 36). Specifically, the definition of BCG unresponsive CIS will also require the following:

  * Pathologically confirmed relapsed or persistent CIS (with or without HG Ta or HG T1 disease) within 12 months of completion (last dose) of adequate BCG treatment for HGUC (e.g., CIS, HG Ta, HG T1, or a combination of these HGUC pathologies).
  * Completion of qualifying BCG treatment (e.g., "5+2" minimum exposure) within 12 months of the initial qualifying dose of BCG (e.g., induction and initial maintenance or re-induction cycle must be completed over no more than a 12-month period of time).
  * Pathological confirmation of BCG unresponsive CIS within 8 weeks of study enrollment.
  * CIS specimen must be predominantly urothelial (transitional cell) and have less than 50% variant (e.g., sarcomatoid, squamous etc. component) histology.
  * No maximum limit to the amount of BCG administered but maintenance BCG should be administered on a schedule consistent with the SWOG 8507 regimen (Lamm 2000).
* Have all Ta and/or T1 disease resected and all CIS resected or fulgurated, as feasible, prior to study treatment (e.g., prior to Day 1 treatment).
* Ineligible to receive radical cystectomy (medically unfit) or refusal of radical cystectomy according to Investigator assessment.
* Demonstrate adequate organ function
* Patients must be willing to comply with study mandated cystoscopies, urine cytology, urograms, biopsies, and other procedures (including TURBT or other resection for all Ta/T1 disease) for the duration of the study. Patients who withdraw consent for these procedures will be withdrawn from the trial

Cohort P Inclusion Criteria

* Be ≥18 years of age (or legal age of majority in the jurisdiction) on day of signing informed consent
* Have ECOG performance status of 0 to 2.
* Have pathologically confirmed (WHO grading system employed for tumor grading) (Compérat 2019) BCG-unresponsive HG Ta/T1 papillary disease without CIS. Patients with BCG-unresponsive HG Ta/T1 papillary disease are those unlikely to benefit from and who will not be receiving further IVE BCG. There is no maximum limit to the amount of prior BCG treatment, but maintenance BCG should be administered on a schedule consistent with standard induction-maintenance protocols. Specifically, the definition of BCG unresponsive HG Ta/T1 papillary disease without CIS will also require the following:

  * Pathologically confirmed recurrent HG Ta/T1 papillary disease without CIS within 6 months of completion (last dose) of adequate BCG treatment for HGUC (e.g., CIS, HG Ta, HG T1, or a combination of these HGUC pathologies).
  * Patients with HG Ta: Completion of qualifying BCG treatment (e.g., "5+2" minimum exposure) within 12 months of the initial qualifying dose of BCG (e.g., induction and initial maintenance or re-induction cycle must be completed over no more than a 12-month period of time).
  * Patients with HG T1: Patients may be eligible after the initial induction alone (5 of 6 doses of an induction course) as the qualifying BCG treatment.
  * Completion (last dose) of qualifying BCG treatment within 12 months of study enrollment.
  * Pathological confirmation of BCG-unresponsive HG Ta/T1 papillary disease without CIS within 14 days of study enrollment.
  * All pathology specimens must be predominantly urothelial (transitional cell) and have less than 50% variant (e.g., sarcomatoid, squamous etc. component) histology.
  * No maximum limit to the amount of BCG administered; however, there should be no more than 12 months between cycles of BCG
* Have all Ta and/or T1 disease resected, prior to study treatment (e.g., prior to Day 1 treatment).
* Ineligible to receive radical cystectomy (medically unfit) or refusal of radical cystectomy based on Investigator assessment.
* Demonstrate adequate organ function,
* Patients must be willing to comply with study-mandated cystoscopies, urine cytology, imaging, biopsies, and other procedures for the duration of the trial

Cohort C and Cohort P Key Exclusion Criteria:

* Has current or past history of muscle invasive (T2 or higher stage) or locally advanced (T3/T4, any N) or metastatic bladder cancer.
* Any HGUC as T1, HG Ta, or CIS in the upper genitourinary tract or prostatic urethra (including CIS of the urethra) within 24 months prior to enrollment OR any history of T2 or higher stage urothelial carcinoma in the upper genitourinary tract (kidneys, renal collecting systems, ureters).
* Has received systemic anti-cancer therapy, including investigational agents, within 4 weeks of Day 1.
* Has had prior systemic treatment (with the exception of checkpoint inhibitor therapy), radiation therapy, or surgery for bladder cancer other than TURBT or bladder biopsies.
* Has any of the following within the 6 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, pulmonary embolus, uncontrolled hypertension, or uncontrolled congestive heart failure.
* Cannot tolerate study-related biopsies, IVE administration, or 1-hour bladder hold of cretostimogene.
* IVE therapy within 8 weeks prior to beginning study treatment with the exception of cytotoxic agents (e.g., Mitomycin C, gemcitabine, doxorubicin and epirubicin) when administered as a single instillation immediately following a TURBT procedure which is permitted 14 or more days prior to beginning study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2027-12-24 (Estimated); Study Completion 2029-12-24 (Estimated)

PRIMARY OUTCOMES:
Cohort C: | 36 months
  To determine the Complete Response rate at any time in patients with BCG-unresponsive CIS with or without concomitant HG Ta/T1 papillary disease.
Cohort P: | 36 months
  To determine the high-grade EFS of cretostimogene in patients with BCG-unresponsive HG Ta/T1 papillary disease without CIS.Ta/T1 papillary disease without CIS.

SECONDARY OUTCOMES:
Cohort C: Duration of response (DOR) | 36 months
  Median duration of response in patients with a CR or PR in subjects
Cohort C and Cohort P: Assess high-grade reoccurrence free survival (RFS) | up to 60 months
Cohort C and Cohort P: Assess progression free survival (PFS ) | up to 60 months
Cohort C:Complete Response rate at 12 months | 12 months
Cohort C and Cohort P : Cystectomy free survival | up to 60 months
Cohort C and Cohort P: Evaluate the safety of Cretostimogene | 36 months
Cohort C: Assess overall survival | up to 60 months
Cohort C: Reoccurrence free survival | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: CG Oncology, Study Director — CG Oncology
Locations (71):
- United States (32):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Arizona Institute of Urology, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - University of California - Irvine, Irvine, California
  - University of Colorado, Aurora, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Urology Associates, Lone Tree, Colorado
  - MedStar Hospital, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Urology of Indiana, Greenwood, Indiana
  - University of Kansas, Kansas City, Kansas
  - Wichita Urology, Wichita, Kansas
  - Southern Urology, Lafayette, Louisiana
  - Chesapeake Urology, Severna Park, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Rochester, Rochester, Minnesota
  - Mercy Medical Center, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Toledo, Toledo, Ohio
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Conrad Pearson Clinic, Germantown, Tennessee
  - Urology Associates- Nashville, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio, PA, San Antonio, Texas
  - Spokane Urology, Spokane, Washington
- Australia (3):
  - Barwon Health, University Hospital Geelong, Geelong
  - Royal Melbourne Hospital, Melbourne
  - Wollongong Private Hospital, Wollongong
- Japan (24):
  - National Cancer Center Hospital East, Chiba
  - Nagoya University Hospital, Fujita
  - Hirosaki University Hospital, Hashimoto
  - Chugoku Rosai Hospital, Hiroshima
  - Shinshu University Hospital, Ishizuka
  - University of Tsukuba Hospital, Kandori
  - Nara Medical University Hospital, Kashihara
  - The Jikei University Kashiwa Hospital, Kashiwa
  - St. Marianna University Hospital, Kikuchi
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Kagawa Rosai Hospital, Marugame
  - Keio University Hospital, Matsumoto
  - Okayama University Hospital, Okayama
  - Osaka City University Hospital, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
  - Kitsato University Hospital, Sagamihara
  - Saitama City Hospital, Saitama
  - Sapporo Medical University Hospital, Sapporo
  - Shizuoka General Hospital, Shizuoka
  - Keio University Hospital, Tokyo
  - Toyoma University Hospital, Toyoma
  - Ehime University Hospital, Tōon
  - Wakayama Medical University Hospital, Wakayama
  - National Hospital Organization Yokohama Medical Center, Yokohama
- South Korea (8):
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang-si
  - Pusan National University Yangsan Hospital, Gyeongsang
  - Chonnam National University Hwasun Hospital, Jeongnam
  - Seoul National University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul
- Taiwan (4):
  - Keelung Chang Gung Memorial Hospital, Keelung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No